CLINICAL TRIAL: NCT06813222
Title: Anemia-Related Outcomes in Patients With CKD Treated With Dapagliflozin
Status: Active, not recruiting | Type: Observational
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Other Study IDs: Dapa-Anemia-DM-CKD
Record Dates: First submitted 2024-09-20; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Anemia; CKD
Keywords: Anemia; CKD; SGLT2i; Dapagliflozin
MeSH Terms: conditions — Anemia | interventions — dapagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Patients with diabetes and CKD receiving Dapagliflozin with and without anemia: Anemia is defined as a baseline of Hb <13.0 g/dl in males and <12.0 g/dl in females
  Interventions: Drug: Dapagliflozin (DAPA)
- Patients with diabetes and CKD receiving antidiabetic drugs other than dapagliflozin: Stable doses of antidiabetic agents (other than dapagliflozin) for ≥4 weeks prior to enrollment.
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — Dapagliflozin 10 mg

SUMMARY:
Anemia-Related Outcomes in Patients with CKD Treated with Dapagliflozin

This study aims to identify factors that predict anemia improvement in chronic kidney disease (CKD) patients using Dapagliflozin, an SGLT2 inhibitor.

Key questions:

* What factors influence how well Dapagliflozin improves anemia in CKD patients?
* Are there specific characteristics that predict better responses to Dapagliflozin treatment?

The investigators will review medical records of CKD patients who started taking Dapagliflozin. The investigators will compare those with low hemoglobin levels (anemia) to those without anemia.

The investigators will analyze:

Changes in hemoglobin levels Other factors related to anemia (e.g., iron levels, TIBC, ferritin) Patient characteristics (e.g., age, sex, CKD stage)

This study will help us understand which CKD patients are most likely to benefit from Dapagliflozin for anemia.

DETAILED DESCRIPTION:
Study Title: Anemia-Related Outcomes in Patients with CKD Treated with Dapagliflozin

Purpose:

This prospective observational study aims to investigate factors associated with anemia improvement in CKD patients treated with Dapagliflozin, a sodium-glucose cotransporter 2 (SGLT2) inhibitor. The study will analyze data from medical records to identify predictors of favorable anemia outcomes in this population.

Study Design:

A prospective cohort study will be conducted using medical records from the Kidney and Urology Center in Alexandria, Egypt. Patients with CKD who initiated Dapagliflozin therapy will be included, and their clinical data will be analyzed to assess the impact of Dapagliflozin on anemia.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 years) diagnosed with CKD based on estimated glomerular filtration rate (eGFR) criteria established by Kidney Disease: Improving Global Outcomes (KDIGO) guidelines.

  * Initiated treatment with Dapagliflozin for a minimum follow-up duration of 12 months.
  * Documented hemoglobin levels before and after Dapagliflozin initiation.
  * For patients receiving antidiabetic drug classes other that Dapagliflozin, they should be on stable doses for at least 4 weeks prior to trial enrollment.
  * For patients treated with ACE inhibitors or ARBs, they should be on stable doses for at least 4 weeks prior to trial enrollment.

Exclusion Criteria:

* • Active malignancy or other life-limiting conditions.

  * Pregnancy.
  * Specific Kidney Diseases: Autosomal dominant or autosomal recessive polycystic kidney disease, Nephrotic syndrome, Lupus nephritis, and ANCA-associated vasculitis.
  * Receiving cytotoxic therapy, immunosuppressive therapy, or other immunotherapy for primary or secondary renal disease within 6 months before enrollment.
  * Receiving therapy with an SGLT2 inhibitors and/or erythropoiesis stimulating agent (ESA) within 8 weeks before enrollment or previous intolerance of an SGLT2 inhibitors.
  * Type 1 diabetes mellitus.
  * Patients who had received red blood cell transfusions within 6 months before enrollment.
  * Patients who had significant active blood loss due to surgical procedures or medical conditions within 12 weeks before, and/or during enrollment.
  * Iron deficiency at baseline defined as a ferritin level <100 ng/mL or a TSAT <20% and a ferritin level 100 to 299 ng/mL.
  * Cause of anemia other than CKD.
  * Patients with Serum iPTH >600 pg/mL at Screening.
  * Receiving any investigational drug within 4 weeks prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The target population for this study consists of adult patients with diabetes chronic kidney disease (CKD) who have initiated treatment with Dapagliflozin, an SGLT2 inhibitor in comparison with patients with diabetes and CKD on antidiabetic drugs other than dapagliflozin
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin Changes | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Amira Kassem, BPharm, MS, PhD, Study Director — Faculty of Pharmacy, Damanhour University, Egypt
Locations (1):
- Damanhour University, Damanhur, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR